CLINICAL TRIAL: NCT04008979
Title: Pharmacokinetic and Pharmacodynamic Assessment of a Novel, Pharmaceutical Lipid-Aspirin Complex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PLx Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 74,290
Record Dates: First submitted 2019-07-02; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Bioequivalence
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: 32 subjects to be randomized to treatment with either immediate release aspirin or PL-ASA at one of two doses (325 mg or 650 mg) administered orally. After completion of the first treatment and a minimum of a two week washout period(14-17 days) subjects are to cross over and receive treatment with the alternative compound at the same dose level.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- PL-ASA 325 mg (Experimental): Novel aspirin formulation being tested
  Interventions: Drug: Aspirin
- IR 325 mg (Active Comparator): Immediate release aspirin
  Interventions: Drug: Aspirin
- PL-ASA-650 (Experimental): Novel aspirin formulation being tested
  Interventions: Drug: Aspirin
- IR 650 (Active Comparator): Immediate release aspirin
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin - lipid complex

SUMMARY:
Prospective, Randomized, Crossover, Bioequivalence study

DETAILED DESCRIPTION:
Active-control crossover study randomizing 32 healthy volunteers to receive one of two dose levels, 325 mg or 650 mg, of either PL-ASA or immediate release aspirin within a two week washout period between treatments. The primary objectives are to assess PK and PD bioequivalence and safety over a twenty four hour period for PL-ASA and immediate release aspirin at 325 mg and 650 mg dose strengths.

ELIGIBILITY:
Inclusion Criteria:

* If female and of childbearing potential, subject has a negative pregnancy test and is not nursing.
* If female and of childbearing potential, subject is using adequate birth control for the duration of the study.
* Subject is able to understand and comply with study procedures.
* Subject is a non-smoker.
* Subject consumes no more than 1 alcoholic drink per day.
* Subject agrees to refrain from alcohol consumption for 48 hours prior to each drug administration and 48 hours after each drug administration.
* Subject is able and willing to provide written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Subject has abnormal screening/baseline laboratory parameters deemed to be clinically significant by the Investigator.
* Subject has taken any prescription medications other than hormone replacement therapy or thyroid replacement hormones within 3 days prior to drug administration.
* Subject has taken any of the following medications within 2 weeks prior to study entry:

  * NSAIDs or other medications for pain, including aspirin or aspirin containing products and acetaminophen (see Appendix B of protocol in Appendix 16.1.1)
  * Proton pump inhibitors, including Prilosec®, Prevacid®, Aciphex®, Protonix®, or Nexium®
  * H-2 blockers, including Tagamet®, Zantac®, Axid®, or Pepcid®
  * Any antiplatelet agent, including Plavix®, Ticlid®, Pletal®, ReoPro®, Integrilin®, Aggrastat®, or Persantine®
  * Any anti-coagulant, including Coumadin®, Acenocoumarol, Phenprocoumon, Phenindione, Heparin, Exanta®, Argatroban, Lepirudin, Hirudin or Bivalirudin
* Subject has used an investigational agent within the past 30 days.
* Subject has hypersensitivity or contraindications to aspirin, ibuprofen, or other NSAID.
* Subject has sensitivity to lecithin.
* Subject has a history of gastrointestinal problems including ulcers, frequent indigestion, or heartburn.
* Subject has a history of stroke, myocardial infarction, or congestive heart failure.
* Subject has a history of asthma, other bronchospastic activity, nasal polyps, or angioedema other than resolved childhood asthma.
* Subject has a history of kidney or liver disease.
* Subject has a history of thrombocytopenia, neutropenia, or bleeding disorder.
* Subject has a history of coronary arterial bypass.
* Subject has a history of non-trauma related hemorrhage.
* Subject has a history of chronic hypertension.
* Subject is currently enrolled in another investigational trial.
* Subject's platelets are unresponsive to arachidonic acid

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2008-02-11 (Actual); Primary Completion 2008-06-10 (Actual); Study Completion 2008-06-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence of PL-ASA and Immediate Release Aspirin AUC0-T | twenty four hours
  Assess for bioequivalence at 325 mg and 650 mg dose levels AUC0-T of the metabolite salicylic acid
Bioequivalence of PL-ASA and Immediate Release Aspirin AUC0-∞ | 24 hours
  Assess for bioequivalence at 325 mg and 650 mg dose levels AUC0-∞ of the metabolite salicylic acid
Bioequivalence of PL-ASA and Immediate Release Aspirin CMAX | 24 hours
  Assess for bioequivalence at 325 mg and 650 mg dose levels CMAX of the metabolite salicylic acid
Bioequivalence of PL-ASA and Immediate Release Aspirin TMAX | 24 hours
  Assess for bioequivalence at 325 mg and 650 mg dose levels TMAX of the metabolite salicylic acid
Bioequivalence of PL-ASA and Immediate Release Aspirin AUC0-24 | 24 hours
  Assess for bioequivalence at 325 mg and 650 mg dose levels AUC0-24 of the percent inhibition of serum Thromboxane B2
Bioequivalence of PL-ASA and Immediate Release Aspirin TMAX STB2 | 24 hours
  Assess for bioequivalence at 325 mg and 650 mg dose levels TMAX of the percent inhibition of serum Thromboxane B2

CONTACTS AND LOCATIONS:
Overall Officials: Upendra Marathi, PhD, Study Director — PLx Pharma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Angiolillo DJ, Bhatt DL, Lanza F, Cryer B, Dong JF, Jeske W, Zimmerman RR, von Chong E, Prats J, Deliargyris EN, Marathi U. Pharmacokinetic/pharmacodynamic assessment of a novel, pharmaceutical lipid-aspirin complex: results of a randomized, crossover, bioequivalence study. J Thromb Thrombolysis. 2019 Nov;48(4):554-562. doi: 10.1007/s11239-019-01933-7. PMID 31420787